CLINICAL TRIAL: NCT01914094
Title: Pre-habilitation Program for Elective Coronary Artery Bypass Graft Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rakesh C. Arora, Medical Director, Intensive Care Cardiac Sciences, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H2010:390
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Patients Waiting for Elective Coronary Artery Bypass Graft Surgery
Keywords: Preoperative care; Exercise therapy; Cardiac surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Received current standard care.
- Prehab (Experimental): Received pre-operative exercise therapy plus education classes concerning management of their risk factors for coronary artery disease at a local medical fitness facility.
  Interventions: Behavioral: Prehab

INTERVENTIONS:
Behavioral: Prehab
  Other Names: Pre-habilitation; Preoperative exercise therapy
  Arms: Prehab

SUMMARY:
Low levels of physical fitness increase the risk of death in patients with cardiovascular disease. Although cardiac rehabilitation programs improve the health of patients after heart surgery, most patients are not referred until after surgery. Therefore, the purpose of this study was to determine if an exercise "pre-habilitation" (i.e., Prehab) program before heart surgery would improve the health of patients before surgery and whether these improvements would be maintained after surgery.

The investigators hypothesized that Prehab would promote the health of patients before heart surgery, and these improvements would be maintained three months post-operatively, as compared to patients who received standard care.

DETAILED DESCRIPTION:
This was a single-centre, parallel randomized controlled trial conducted in Canada to determine the feasibility and efficacy of an exercise and education "pre-habilitation" (i.e., Prehab) program before elective coronary artery bypass graft surgery (CABG). We recruited 17 patients who were scheduled to undergo elective CABG surgery from February 2011-May 2012. Enrolled patients were assessed at baseline, one week pre-operatively, and three months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* On elective waitlist for coronary artery bypass graft surgery with a minimum anticipated wait time of 4-6 weeks or more
* No history of unstable angina
* Canadian Cardiovascular Society score of less than 4
* No history of myocardial infarction within the past 7 days
* Ejection fraction greater than 30%
* No history of dementia or psychiatric problems
* No self-reported dizziness or confusion
* Able to read, speak, and understand English
* Previously sedentary (reporting accumulating less than 45 minutes of moderate intensity physical activity per day on at least three days per week over the last three months)
* No previous participation in cardiac rehabilitation
* Lives in Winnipeg, Manitoba, Canada or has easy access to the Reh-Fit Centre (local medical fitness facility)

Exclusion Criteria:

* If patients cannot attend Prehab due to geographical limitations
* If patients cannot participate due to physical limitations
* Diagnosis of exercise-induced arrhythmia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walking distance | Baseline; 1 week pre-operatively; 3 months post-operatively
  Assessed using the 6-minute walking test. Output is distance. Change from baseline 6-minute walking distance was assessed at each follow-up time point.

SECONDARY OUTCOMES:
Change in 5-meter gait speed | Baseline; 1 week pre-operatively; 3 months post-operatively
  Assessed using the 5-meter gait speed test. Output is seconds. Change from baseline 5-meter gait speed was assessed at each follow-up time point.
Change in objectively measured physical activity | Baseline; 1 week pre-operatively; 3 months post-operatively
  Measured by accelerometry. Output is minutes of moderate-vigorous as well as total physical activity per week. Change from baseline physical activity was assessed at each follow-up time point.
Change in quality of life | Baseline; 1 week pre-operatively; 3 months post-operatively
  Self-reported using the Short Form-36 questionnaire. Output is a summary score across eight dimensions: General health, Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/fatigue, Pain, Emotional well-being, and Social functioning. Change from baseline quality of life measures was assessed at each follow-up time point.
Change in depressive symptoms | Baseline; 1 week pre-operatively; 3 months post-operatively
  Assessed using the Patient Health Questionnaire-9. Output was a numerical and categorical score. Change from baseline depressive symptoms was assessed at each follow-up time point.
Change in exercise self-efficacy | Baseline; 1 week pre-operatively; 3 months post-operatively
  Assessed by the Cardiac Exercise Self-efficacy Index. Output was a numerical score. Change from baseline exercise self-efficacy was assessed at each follow-up time point.
Change in cardiac anxiety | Baseline; 1 week pre-operatively; 3 months post-operatively
  Assessed by the Cardiac Anxiety Questionnaire. Outputs were numerical scores across four dimensions: Fear, Avoidance, Heart-Focused Attention, and Total Score. Change from baseline cardiac anxiety was assessed at each follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Ann V Sawatzky, PhD, Principal Investigator — University of Manitoba; Rakesh C Arora, MD, Principal Investigator — University of Manitoba
Locations (1):
- Reh-Fit Centre, Winnipeg, Manitoba, Canada